CLINICAL TRIAL: NCT04713267
Title: ISABel: Intelligent Sleep Apnoea Bed
Acronym: ISABel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting participants
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: ISABel Bed 1 and ISABel Bed 2
Record Dates: First submitted 2020-12-17; First posted 2021-01-19 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Effect of ISABel Bed 1 Ans ISABel Bed 2
Keywords: Effect; Comparation; User Feasibility; Tolerance

STUDY DESIGN:
Intervention Model Description: Randomised crossover interventional trial allocating patients with POSA to ISABel Bed 1 or ISABel Bed 2 in random order to study the effect on POSA. Patients with POSA (untreated, or if treated, following a short-term therapy withdrawal) will undergo an in-laboratory polysomnography in ISABel Bed 1 and Bed 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ISABel Bed 1 or ISABel Bed 2 (Other): The study has a within-subject repeated measures-design. After a baseline measurement, participants will be allocated to either a first experimental night in automated bed 1 (ISABel Bed 1) and a second one in automated bed 2 (ISABel Bed 2) or a first experimental night in bed 2 and a second one in bed 1. Afterwards, the results of each polysomnographic measurement carried out during the intervention will be compared to the off-treatment baseline measurement.
  Interventions: Device: ISABel Bed 1

INTERVENTIONS:
Device: ISABel Bed 1 — During the intervention nights (2 out of 3 experiment nights), positional therapy by means of the automated bed will be applied in order to induce a change in the sleeping position.

SUMMARY:
The aim of this trial is to assess the effect of two automated beds on severity of POSA as well as the feasibility of these beds as POSA treatment. These beds are equipped with sensors detecting apnoeas and hypopnoeas from physiological measurements - such as chest movement or breathing sound -, and coherently reacting by actively changing the user position whenever an apnoeic event occurs. Thereby we will investigate a possible treatment alternative to already established OSA therapies, either as a valuable add-on for patients eligible to the currently available therapies or as primary treatment option.

DETAILED DESCRIPTION:
During the intervention nights (2 out of 3 experiment nights), positional therapy by means of the automated bed will be applied in order to induce a change in the sleeping position. Two approaches to influence the position will be investigated:

1. Lifting the upper body up, which has been suggested as a method for reducing habitual snoring. This intervention will be provided by an adjustable bed (AmbianceE-Motion, manufactured by Elite SA, Aubonne, Switzerland) referred to as ISABel Bed 1. This bed contains four motors for changing the inclination angle of the head, trunk, leg, and foot support. Only the position of the trunk and head support is changed during the study. The inclination angle is set to the maximum inclination angle the bed allows: this is 50° at the slatted frame which results in approximately 40° inclination of the hip of the user. The reference angle (0°) is represented by the supine position.
2. Inclination of one side of the bed. This intervention will be provided with a custom-made, adjustable bed base prototype, referred to as ISABel Bed 2 (produced by Sensory-Motor Systems Lab, ETH Zurich, Zurich, Switzerland). The bed is equipped with two motors which allow sideward inclination of up to 40 °. The inclination to be applied in this study is set to 30 ° based on a pre-study with healthy human subjects. Both beds are equipped with non-invasive, cable-free sensors (cardio-ballistography, microphone, and force sensor). A closed-loop control algorithm, which has been developed using machine learning techniques, continuously monitors these signals and triggers the positional intervention, when it detects that the participant is experiencing an apnoea event.

ELIGIBILITY:
Inclusion Criteria:

* Documented supine positional OSA (AHIsupine/AHInonsupine ≥2) with a total AHI of ≥10 events/hour
* Age ≥18 years and <80 years
* Written informed consent documented by signature

Exclusion Criteria:

* Previous or current use of positional therapy
* Use of home oxygen therapy
* Documented hypoventilation syndrome
* Documented Cheyne-Stokes breathing
* Documented moderate-to-severe or severe obstructive lung diseases
* Chronic heart failure
* Documented active drug or alcohol abuse
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, documented psychological disorders, documented dementia, etc. of the participant
* Current professional driver or any either documented or reported previous sleep-related driving accidents
* People working with or operating heavy machinery
* Child-bearing age: female participants who are neither surgically sterilised / hysterectomised nor post-menopausal for longer than 2 years are considered as being of child bearing potential
* Documented unstable, untreated coronary or peripheral artery disease, severe hypertension or hypotension (≥180/110 or ≤90/60 mmHg)
* BMI >40 kg/m2 or body weight >130 kg
* Being the investigator, his/her family members, employees, or other dependent persons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Assessment of the presence of a difference in supine AHI either in ISABel Bed 1 or ISABel Bed 2 | three nights
  The primary outcome will be the presence of a difference in supine AHI (events/hour) between the control bed (polysomnography - PSG- on Day 6) and either ISABel Bed 1 or ISABel Bed 2 (respectively on Day 7 and Day 8 to 14, depending on the randomisation order). AHI supine refers to the part of the total AHI that is caused by lying in supine position. This index is per definition twice as much as the non-supine AHI in patients with POSA. The intervention should reduce the time spent in supine position and therefore reduce the supine AHI.

SECONDARY OUTCOMES:
User feasibility of ISABel Bed 1 or ISABel Bed 2 | three nights
  snoring, sleep architecture
User effect of ISABel Bed 1 or ISABel Bed 2 | three nights
  total AHI (events/hours), ODI4%, SpO2%, total arousal index (events/hours)
User tolerance | three nights
  morning blood pressure and heart rate
Difference ISABel Bed 1 and ISABel Bed 2 | three nights
  in supine AHI between the two beds
Assess reliability fo the machine learning algorithms of ISABel Bed 1 and ISABel Bed 2 | three nights
  data collection
Safety of ISABel Bed 1 and ISABel Bed 2 | three nights
  Sleep structure and quality

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland